CLINICAL TRIAL: NCT05608850
Title: Acute Responses of Postural Alignment, Kinematic Synergy, and Intermuscular Coherence to Postural Muscle Facilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radford University (Other)
Responsible Party: Principal Investigator, Stephen Glass, Assistant Professor, Radford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-288-RUC
Record Dates: First submitted 2022-10-28; First posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Posture; Musculoskeletal Equilibrium; Electromyography; Kinematics
Keywords: Alignment; Posture; Motor control; Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Then Stretch (Other): Participants in AB will perform the experimental (exercise) intervention first and the control (stretch) intervention second
  Interventions: Other: Exercise Then Stretch; Other: Stretch Then Exercise
- Stretch Then Exercise (Other): Participants in BA will perform the experimental (exercise) intervention second and the control (stretch) intervention first
  Interventions: Other: Exercise Then Stretch; Other: Stretch Then Exercise

INTERVENTIONS:
Other: Exercise Then Stretch — This arm (sequence) will perform an anti-gravity kinetic chain intervention and then a passive, partner-assisted stretching intervention, separated by a one-week washout period.
Other: Stretch Then Exercise — This arm (sequence) will perform a passive, partner-assisted stretching intervention and then an anti-gravity kinetic chain intervention , separated by a one-week washout period.

SUMMARY:
Clinicians frequently assess and intervene on postural alignment. However, research demonstrating the effects of exercise interventions in moving postural alignment toward an evidence-based standard is lacking. Part of the difficulty in establishing such evidence has been a lack of theory-motivated conceptions of what "good" posture is. In other words, the prevailing understanding of postural alignment is based on the negation of what has been observed to associate with bad outcomes. This study will build upon preliminary findings from our laboratory that define good postural alignment on theoretical grounds. The investigators will measure motion capture and muscle activation patterns during simple postural alignment tasks before and after 1) a corrective exercise intervention, or 2) a control intervention based designed to inhibit superficial muscle tension. The corrective exercise intervention is designed to counteract the natural patterns in which the human skeleton tends to collapse from a standing position under the influence of gravity. The control intervention consists of passive, partner-assisted stretching. Regardless of initial assignment, all participants will crossover (i.e. switch interventions) and repeat the study procedures after a 1-week washout period. Behavioral indicators of movement and nervous system coordination will be used to quantify alignment before and after exercise, as well as the consistency of those alignment patterns with theoretically-defined standards. The knowledge gained from this study will contribute to evidence-based definitions of healthy postural alignment and help identify effective interventions by which clinicians can promote good posture.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* 18 - 40 years of age

Exclusion Criteria:

* Recent (< 6 months) history of lower extremity injury
* Recent (< 6 months) history of other musculoskeletal or neurological disorder affecting balance
* Contraindications to participation in physical activity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Euclidean distance from the vector describing subject-specific, simulated gravitational collapse | Immediately before Intervention (Day 1)
  This outcome is a cumulative descriptor of segment angle distance from the pattern in which an individual's posture would collapse. The reference point for each individual is calculated using both pre and post-intervention data for a given day.
Euclidean distance from the vector describing subject-specific, simulated gravitational collapse | Immediately after Intervention (Day 1)
  This outcome is a cumulative descriptor of segment angle distance from the pattern in which an individual's posture would collapse. The reference point for each individual is calculated using both pre and post-intervention data for a given day.
Euclidean distance from the vector describing subject-specific, simulated gravitational collapse | Immediately before Intervention (Day 7)
  This outcome is a cumulative descriptor of segment angle distance from the pattern in which an individual's posture would collapse. The reference point for each individual is calculated using both pre and post-intervention data for a given day.
Euclidean distance from the vector describing subject-specific, simulated gravitational collapse | Immediately after Intervention (Day 7)
  This outcome is a cumulative descriptor of segment angle distance from the pattern in which an individual's posture would collapse. The reference point for each individual is calculated using both pre and post-intervention data for a given day.
Pooled intermuscular coherence | Immediately before Intervention (Day 1)
  Weighted average of frequency-domain correlations between muscle pairs belonging to anterior, posterior, and trunk muscle groups.
Pooled intermuscular coherence | Immediately after Intervention (Day 1)
  Weighted average of frequency-domain correlations between muscle pairs belonging to anterior, posterior, and trunk muscle groups.
Pooled intermuscular coherence | Immediately before Intervention (Day 7)
  Weighted average of frequency-domain correlations between muscle pairs belonging to anterior, posterior, and trunk muscle groups.
Pooled intermuscular coherence | Immediately after Intervention (Day 7)
  Weighted average of frequency-domain correlations between muscle pairs belonging to anterior, posterior, and trunk muscle groups.

SECONDARY OUTCOMES:
Top-down kinetic chain continuity | Immediately before Intervention (Day 1)
  The purpose of this outcome is to quantify the communication of motion from the upper body to the lower body. In a test involving placing hands-on-head and pulling the elbows back as far as possible, the response in the lower body is quantified by posterior rotation of the tibial segment.
Top-down kinetic chain continuity | Immediately after Intervention (Day 1)
  The purpose of this outcome is to quantify the communication of motion from the upper body to the lower body. In a test involving placing hands-on-head and pulling the elbows back as far as possible, the response in the lower body is quantified by posterior rotation of the tibial segment.
Top-down kinetic chain continuity | Immediately before Intervention (Day 7)
  The purpose of this outcome is to quantify the communication of motion from the upper body to the lower body. In a test involving placing hands-on-head and pulling the elbows back as far as possible, the response in the lower body is quantified by posterior rotation of the tibial segment.
Top-down kinetic chain continuity | Immediately after Intervention (Day 7)
  The purpose of this outcome is to quantify the communication of motion from the upper body to the lower body. In a test involving placing hands-on-head and pulling the elbows back as far as possible, the response in the lower body is quantified by posterior rotation of the tibial segment.

CONTACTS AND LOCATIONS:
Locations (1):
- Radford University Carilion, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data for individual participants will be shared upon request with parties committing to institutional data sharing agreements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: On request and indefinitely.